CLINICAL TRIAL: NCT04716361
Title: Clinical and Economic Outcome of Endovascular Therapies in Chronic Femoropopliteal Occlusive Disease With Severe Calcification (The Evolution Study): a Prospective, Multi-center，Observational Study
Brief Title: Outcome of Endovascular Therapies in Chronic Femoropopliteal Occlusive Disease With Severe Calcification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20200011B
Record Dates: First submitted 2021-01-10; First posted 2021-01-20 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Femoropopliteal Artery Occlusion
Keywords: Peripheral artery disease; Calcification; Endovascular treatment
MeSH Terms: conditions — Peripheral Arterial Disease; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, multicenter, real world, observational study, which aims at evaluating the safety, efficacy and economic cost of endovascular treatments for endovascular therapies in chronic femoropopliteal occlusive disease with severe calcification. It is estimated that 400 subjects diagnosed with chronic femoropopliteal occlusive disease with severe calcification and receive endovascular treatments will be enrolled in eight centers nationwide from January 2021 to December 2022. All the subjects will be under follow-up for two years. There is no restriction on the endovascular techniques. The primary outcomes include the technical success rate of each endovascular techniques and the reintervention rate driven by lesions' clinical symptoms.

DETAILED DESCRIPTION:
Arteriosclerosis obliterans (ASO) is a common disease in middle-aged and elderly people, which affects up to 30% people who are over 70 years in the general population. Its symptoms include claudication, rest pain and ischemic tissue loss depending on its severity. Nowadays, endovascular treatments have become the first-line therapy. If ASO is combined with severe calcification, the treatment will be much more challenging. The efficacy of plain old balloon angioplasty is limited. New devices including drug-coated balloon, intravascular Lithotripsy, directional atherectomy, Supera stent and drug-eluting stent offer another chance and better prognosis. The data of these new devices, however, are mainly from low quality evidence. Therefore, we start this prospective, multicenter, real world, observational study, providing new data on the safety, efficacy and health economics evaluation of endovascular treatments for endovascular therapies in chronic femoropopliteal occlusive disease with severe calcification.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford stages 2-6
2. The target vessel (femoral and/or popliteal artery) has at least ≥90% stenosis or occlusion with the moderate to severe calcification (defined as >5 cm continuous calcification)
3. For patients with both lower limbs to be treated, the side with severer calcification is selected. If the calcification is similar in the two sides, the first one to be treated is selected.
4. At least one outflow artery (which is patent in > 1/3 length) in the calf connects the popliteal artery.
5. Patients who failed the first treatment because the guide wire could not pass through the lesion can still be selected if the second endovascular treatment succeeds.
6. There is no restriction on the types of endovascular techniques and devices.

Exclusion Criteria:

Exclusion Criteria:

1. Life expectation less than one year
2. There is several infection and/or major tissue loss in the leg. Even if after revascularization, patient still need amputation.
3. The quality of patients' life cannot be assessed by vascular quality of life questionnaire due to difficulties in communication.
4. Chronic femoropopliteal occlusive disease without calcification.
5. Patients with acute arterial thrombosis.
6. Limbs that have been treated with the femoral and popliteal artery bypass surgery.
7. Pregnant women
8. Allergic to contrast medium
9. Participating in other drug or device studies currently.
10. Systematic infection and/or coagulation disorders 14 days before the enrollment.
11. Patients have severe systematic disease that cannot be controlled currently such as severe heart, lung disease, live function disorder, end stage cancer, etc
12. Stroke, myocardial infarction, bleeding in the past 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic femoropopliteal occlusive disease with severe calcification
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 1 week
  Successfully revascularize the target vessel. The residual stenosis is <30% and there is no acute thrombosis occurred in the target vessel within 1 week post-operation.
The clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 1 month
  Any reintervention within the target lesion due to symptoms or drop of ≥20% ABI compared to baseline.
The clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 6 months
  Any reintervention within the target lesion due to symptoms or drop of ≥20% ABI compared to baseline.
The clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 12 months
  Any reintervention within the target lesion due to symptoms or drop of ≥20% ABI compared to baseline.
The clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 18 months
  Any reintervention within the target lesion due to symptoms or drop of ≥20% ABI compared to baseline.
The clinically driven target lesion revascularization(CD-TLR) rate at post-interventional | 24 months
  Any reintervention within the target lesion due to symptoms or drop of ≥20% ABI compared to baseline.

SECONDARY OUTCOMES:
Vascular quality of life questionnaire(VascuQol) | 1 month,6 months,12 months,18 months and 24 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Incidence of severe adverse events | 1 month,6 months,12 months,18 months and 24 months
  Severe adverse events include anyone of the following: Myocardial infarction, ischemic stroke, cardiovascular mortality, acute limb ischemia, and major amputation of a vascular etiology.
Patency of the target vessel | Patency of the target vessel. [ Time Frame: 1 month,6 months,12 months,18 months and 24 months
  The patency is assessed by the vascular ultrasound.
Health economics evaluation | 24 months
  All the cost related to the target vessel and spent in the inpatient ward will be recorded and analyzed.
Wound, Ischemia, and foot infection(WIFI) classification system | 1 month,6 months,12 months,18 months and 24 months
  The Wound, Ischemia, and foot Infection (WIfI) classification system is a composite outcome measure encompassing demographic changes and expanding techniques of revascularization to perform meaningful analyses of outcomes in the treatment of the threatened limb, including wound, ischemia and foot infection. Each index was evaluated by very low, low, moderate and high, the very low represents no risk, the high reveals high risk of amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Ziheng Wu, M.D., Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Dua A, Lee CJ. Epidemiology of Peripheral Arterial Disease and Critical Limb Ischemia. Tech Vasc Interv Radiol. 2016 Jun;19(2):91-5. doi: 10.1053/j.tvir.2016.04.001. Epub 2016 Apr 22. PMID 27423989
- [Background] Olinic DM, Spinu M, Olinic M, Homorodean C, Tataru DA, Liew A, Schernthaner GH, Stanek A, Fowkes G, Catalano M. Epidemiology of peripheral artery disease in Europe: VAS Educational Paper. Int Angiol. 2018 Aug;37(4):327-334. doi: 10.23736/S0392-9590.18.03996-2. PMID 29936722
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] Rocha-Singh KJ, Zeller T, Jaff MR. Peripheral arterial calcification: prevalence, mechanism, detection, and clinical implications. Catheter Cardiovasc Interv. 2014 May 1;83(6):E212-20. doi: 10.1002/ccd.25387. Epub 2014 Feb 10. PMID 24402839
- [Background] Okuno S, Iida O, Shiraki T, Fujita M, Masuda M, Okamoto S, Ishihara T, Nanto K, Kanda T, Takahara M, Uematsu M. Impact of Calcification on Clinical Outcomes After Endovascular Therapy for Superficial Femoral Artery Disease: Assessment Using the Peripheral Artery Calcification Scoring System. J Endovasc Ther. 2016 Oct;23(5):731-7. doi: 10.1177/1526602816656612. Epub 2016 Jul 1. PMID 27369975
- [Background] He HP, Weng JC, Zhao Y, Cai SH, Zhang XL, Yin HH. Impact of Plaque Calcification and Stent Oversizing on Clinical Outcomes of Atherosclerotic Femoropopliteal Arterial Occlusive Disease Following Stent Angioplasty. Eur J Vasc Endovasc Surg. 2019 Aug;58(2):215-222. doi: 10.1016/j.ejvs.2019.01.025. Epub 2019 Mar 9. PMID 30862415
- [Background] Tepe G, Beschorner U, Ruether C, Fischer I, Pfaffinger P, Noory E, Zeller T. Drug-Eluting Balloon Therapy for Femoropopliteal Occlusive Disease: Predictors of Outcome With a Special Emphasis on Calcium. J Endovasc Ther. 2015 Oct;22(5):727-33. doi: 10.1177/1526602815600156. Epub 2015 Aug 6. PMID 26250747
- [Background] Cassese S, Wolf F, Ingwersen M, Kinstner CM, Fusaro M, Ndrepepa G, Ibrahim T, Ott I, Lammer J, Krankenberg H, Fusaro M. Drug-Coated Balloon Angioplasty for Femoropopliteal In-Stent Restenosis. Circ Cardiovasc Interv. 2018 Dec;11(12):e007055. doi: 10.1161/CIRCINTERVENTIONS.118.007055. PMID 30562083
- [Background] Chen Z, Guo W, Jiang W, Wang F, Fu W, Zou Y, Deckers S, Li P, Popma JJ, Jaff MR. IN.PACT SFA Clinical Study Using the IN.PACT Admiral Drug-Coated Balloon in a Chinese Patient Population. J Endovasc Ther. 2019 Aug;26(4):471-478. doi: 10.1177/1526602819852084. Epub 2019 Jun 17. PMID 31204595
- [Background] Caradu C, Lakhlifi E, Colacchio EC, Midy D, Berard X, Poirier M, Ducasse E. Systematic review and updated meta-analysis of the use of drug-coated balloon angioplasty versus plain old balloon angioplasty for femoropopliteal arterial disease. J Vasc Surg. 2019 Sep;70(3):981-995.e10. doi: 10.1016/j.jvs.2019.01.080. Epub 2019 May 21. PMID 31126769
- [Background] Brodmann M, Schwindt A, Argyriou A, Gammon R. Safety and Feasibility of Intravascular Lithotripsy for Treatment of Common Femoral Artery Stenoses. J Endovasc Ther. 2019 Jun;26(3):283-287. doi: 10.1177/1526602819844998. Epub 2019 Apr 22. PMID 31006305
- [Background] Adams G, Shammas N, Mangalmurti S, Bernardo NL, Miller WE, Soukas PA, Parikh SA, Armstrong EJ, Tepe G, Lansky A, Gray WA. Intravascular Lithotripsy for Treatment of Calcified Lower Extremity Arterial Stenosis: Initial Analysis of the Disrupt PAD III Study. J Endovasc Ther. 2020 Jun;27(3):473-480. doi: 10.1177/1526602820914598. Epub 2020 Apr 3. PMID 32242768
- [Background] Bohme T, Romano L, Macharzina RR, Noory E, Beschorner U, Jacques B, Burgelin K, Flugel PC, Zeller T, Rastan A. Outcomes of directional atherectomy for common femoral artery disease. EuroIntervention. 2021 Jun 25;17(3):260-266. doi: 10.4244/EIJ-D-19-00693. PMID 32176618
- [Background] Bisdas T, Beropoulis E, Argyriou A, Torsello G, Stavroulakis K. 1-Year All-Comers Analysis of the Eluvia Drug-Eluting Stent for Long Femoropopliteal Lesions After Suboptimal Angioplasty. JACC Cardiovasc Interv. 2018 May 28;11(10):957-966. doi: 10.1016/j.jcin.2018.03.046. PMID 29798772
- [Background] Cioppa A, Stabile E, Salemme L, Popusoi G, Pucciarelli A, Iacovelli F, Arcari A, Coscioni E, Trimarco B, Esposito G, Tesorio T. Combined use of directional atherectomy and drug-coated balloon for the endovascular treatment of common femoral artery disease: immediate and one-year outcomes. EuroIntervention. 2017 Feb 20;12(14):1789-1794. doi: 10.4244/EIJ-D-15-00187. PMID 28216476
- [Background] Mohapatra A, Saadeddin Z, Bertges DJ, Madigan MC, Al-Khoury GE, Makaroun MS, Eslami MH. Nationwide trends in drug-coated balloon and drug-eluting stent utilization in the femoropopliteal arteries. J Vasc Surg. 2020 Feb;71(2):560-566. doi: 10.1016/j.jvs.2019.05.034. Epub 2019 Aug 10. PMID 31405761
- [Background] Stavroulakis K, Schwindt A, Torsello G, Beropoulis E, Stachmann A, Hericks C, Bollenberg L, Bisdas T. Directional Atherectomy With Antirestenotic Therapy vs Drug-Coated Balloon Angioplasty Alone for Common Femoral Artery Atherosclerotic Disease. J Endovasc Ther. 2018 Feb;25(1):92-99. doi: 10.1177/1526602817748319. Epub 2017 Dec 18. PMID 29251204
- [Background] Kokkinidis DG, Jawaid O, Cantu D, Martinsen BJ, Igyarto Z, Valle JA, Waldo SW, Armstrong EJ. Two-Year Outcomes of Orbital Atherectomy Combined With Drug-Coated Balloon Angioplasty for Treatment of Heavily Calcified Femoropopliteal Lesions. J Endovasc Ther. 2020 Jun;27(3):492-501. doi: 10.1177/1526602820915244. Epub 2020 May 4. PMID 32364000
- [Derived] Wang B, Xu Y, Yu X, Sun S, Guo L, Ye M, He C, Li Q, Feng Z, Wu Z. Endovascular Treatment for Calcified Femoropopliteal Peripheral Artery Disease and Risk Factor Identification: Two Year Outcomes of the Evolusion Study. Eur J Vasc Endovasc Surg. 2025 Oct 4:S1078-5884(25)01001-9. doi: 10.1016/j.ejvs.2025.10.002. Online ahead of print. PMID 41052588
- [Derived] Pan J, Guo L, Fang X, Feng Z, Li Q, He C, Sang H, Shi W, Shi Z, Wang B, Qiu C, Wu Z, Ye M. Protocol of the evolution study: A prospective, multicenter, observational study evaluating the effect and health economics of endovascular treatment in patients with moderate and severe calcification of femoropopliteal artery. Front Cardiovasc Med. 2022 Oct 18;9:1039313. doi: 10.3389/fcvm.2022.1039313. eCollection 2022. PMID 36330013